CLINICAL TRIAL: NCT00489554
Title: Primary Vaccination Course in Children Receiving the Pneumococcal Vaccine GSK 1024850A, Infanrix Hexa and Rotarix
Brief Title: Primary Vaccination Study With a Pneumococcal Conjugate Vaccine in Healthy Children 6 to 12wks of Age
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 109661; 2015-001510-10 (EudraCT Number)
Record Dates: First submitted 2007-06-20; First posted 2007-06-21 (Estimated); Results first posted 2012-05-10 (Estimated); Last update posted 2020-01-13 (Actual); Status verified 2019-12

CONDITIONS: Infections, Streptococcal; Streptococcus Pneumoniae Vaccines
Keywords: Primary vaccination; Safety; Pneumococcal vaccine.; Pneumococcal disease; Immunogenicity
MeSH Terms: conditions — Streptococcal Infections; Pneumococcal Infections | interventions — PHiD-CV vaccine; diphtheria-tetanus-acellular pertussis-inactivated poliovirus-Haemophilus influenzae b conjugate-hepatitis B vaccine; RIX4414 vaccine

ARMS (1):
- Synflorix Vaccine Group (Experimental): Subjects receiving Synflorix vaccine co-administered with DTPa-HBV-IPV/Hib (Infanrix hexa) vaccine at 2-4-6 months of age, and co-administered with HRV (Rotarix) vaccine at 2-4 months of age.
  Interventions: Biological: Synflorix; Biological: Infanrix hexa; Biological: Rotarix

INTERVENTIONS:
Biological: Synflorix — Intramuscular injection, 3 doses.
  Other Names: Pneumococcal conjugate vaccine GSK1024850A.
Biological: Infanrix hexa — Intramuscular injection, 3 doses.
Biological: Rotarix — Oral, 2 doses.

SUMMARY:
The purpose of this study is to assess the immunogenicity in terms of antibody response and the safety/reactogenicity in terms of solicited and unsolicited symptoms and serious adverse events following primary vaccination of Mexican infants with pneumococcal conjugate vaccine GSK 1024850A co-administered with a diphtheria, tetanus, acellular pertussis (DTPa)-combined vaccine (Infanrix hexa) and rotavirus vaccine (Rotarix) in children during the first 6 months of age.

DETAILED DESCRIPTION:
The Protocol Posting has been updated in order to comply with the FDA Amendment Act, Sep 2007.

ELIGIBILITY:
Inclusion Criteria:

* Male or female subjects between and including 6-12 weeks of age at the time of the first vaccination.
* Subjects for whom the investigator believes that their parents/guardians can and will comply with the requirements of the protocol.
* Written informed consent obtained from the parent or guardian of the subject.
* Free of obvious health problems as established by medical history and clinical examination before entering into the study.
* Born after a gestation period of 36 to 42 weeks inclusive.

Exclusion Criteria:

* Use of any investigational or non-registered product (drug or vaccine) other than the study vaccine(s) within 30 days preceding the first dose of study vaccine, or planned use during the study period.
* Planned administration/administration of a vaccine not foreseen by the study protocol during the period starting one month before each dose of vaccines and ending 7 days after dose 1 and dose 2 and one month after dose 3.
* Concurrently participating in another clinical study, at any time during the study period, in which the subject has been or will be exposed to an investigational or a non-investigational product.
* Chronic administration (defined as more than 14 days) of immunosuppressants or other immune-modifying drugs since birth.
* A family history of congenital or hereditary immunodeficiency.
* Any confirmed or suspected immunosuppressive or immunodeficient condition based on medical history and physical examination.
* Administration of immunoglobulins and/or any blood products since birth or planned administration during the study period.
* Previous vaccination against diphtheria, tetanus, pertussis, polio, hepatitis B, Haemophilus influenzae type b, rotavirus and/or Streptococcus pneumoniae; with the exception of vaccines where the first dose may be given at birth within the first two weeks of life according to national recommendations (e.g. Hepatitis B and BCG).
* History of, or intercurrent, diphtheria, tetanus, pertussis, polio, hepatitis B and Haemophilus influenzae type b disease.
* Gastroenteritis within 7 days preceding the study vaccine administration (warrants deferral of the vaccination).
* Any clinically significant history of chronic gastrointestinal disease including any uncorrected congenital malformation of the gastrointestinal (GI) tract, intussusception (IS) or other medical condition determined to be serious by the investigator.
* History of allergic disease or reactions likely to be exacerbated by any component of the vaccines.
* History of any neurological disorders or seizures.
* Major congenital defects or serious chronic illness.
* Acute disease at the time of enrolment.

Ages: 6 Weeks to 12 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 230 (Actual)
Dates: Start 2007-07-03 (Actual); Primary Completion 2008-03-31 (Actual); Study Completion 2008-03-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline
Locations (2):
- Mexico (2):
  - GSK Investigational Site, Mexico City
  - GSK Investigational Site, México

IPD SHARING:
Plan to Share IPD: Yes
IPD is available via the Clinical Study Data Request site (click on the link provided below).
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: IPD is available via the Clinical Study Data Request site (click on the link provided below).
Access Criteria: Access is provided after a research proposal is submitted and has received approval from the Independent Review Panel and after a Data Sharing Agreement is in place. Access is provided for an initial period of 12 months but an extension can be granted, when justified, for up to another 12 months.
URL: https://clinicalstudydatarequest.com/Posting.aspx?ID=256

REFERENCES:
- [Background] Ruiz-Palacios G et al. Immunogenicity, safety and reactogenicity of the new 10-valent pneumococcal non-typeable Haemophilus influenzae protein D-conjugate vaccine (PHiD-CV) in Mexican infants. Abstract presented at the XIII Congreso Latinoamericano de Infectología Pediátrica (SLIPE). Guayaquil, Ecuador, 12-15 August 2009.
- [Background] Ruiz-Palacios GM, Guerrero ML, Hernandez-Delgado L, Lavalle-Villalobos A, Casas-Munoz A, Cervantes-Apolinar Y, Moreira M, Schuerman L. Immunogenicity, reactogenicity and safety of the 10-valent pneumococcal nontypeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV) in Mexican infants. Hum Vaccin. 2011 Nov;7(11):1137-45. doi: 10.4161/hv.7.11.17984. Epub 2011 Nov 1. PMID 22048109
- [Background] Schuerman L et al. Population variability in antibody responses following pneumococcal conjugate vaccination: experience with the non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV). Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- [Background] Schuerman L et al. Population variability of opsonophagocytic activity following 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate (PHiD-CV) vaccination more limited than antibody responses. Abstract presented at the 7th International Symposium on Pneumococci and Pneumococcal Diseases (ISPPD). Tel Aviv, Israel, 14-18 March 2010.
- [Background] Silfverdal SA, Coremans V, Francois N, Borys D, Cleerbout J. Safety profile of the 10-valent pneumococcal non-typeable Haemophilus influenzae protein D conjugate vaccine (PHiD-CV). Expert Rev Vaccines. 2017 Feb;16(2):109-121. doi: 10.1586/14760584.2016.1164044. Epub 2016 Sep 30. PMID 26954689
- See also: Researchers can use this site to request access to anonymised patient level data and/or supporting documents from clinical studies to conduct further research. — https://www.clinicalstudydatarequest.com
- Available data/document: Statistical Analysis Plan: 109661 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Individual Participant Data Set: 109661 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Dataset Specification: 109661 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Clinical Study Report: 109661 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Informed Consent Form: 109661 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register
- Available data/document: Study Protocol: 109661 — https://www.clinicalstudydatarequest.com — For additional information about this study please refer to the GSK Clinical Study Register

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Synflorix Vaccine Group
Started | 230
Completed | 226
Not Completed | 4
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 1

BASELINE CHARACTERISTICS:
Arm/Group | Synflorix Vaccine Group
Number analyzed (Participants) | 230
Age, Continuous [Mean (Standard Deviation); unit: weeks] | 8.2 (1.63)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 123
  Male | 107

OUTCOME MEASURES:

1. Primary Outcome: Antibody Concentrations Against Pneumococcal Vaccine Serotypes
Description: Concentrations were expressed as geometric mean concentration (GMC). The vaccine pneumococcal serotypes assessed include 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F, and 23F.
Time Frame: One month after the administration of the 3rd vaccine dose i.e. Month 5
Population: Analysis was performed on According-to-Protocol (ATP) cohort for immunogenicity which included all evaluable subjects for whom immunogenicity data were available.
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter
Arm/Group | Synflorix Vaccine Group
Number analyzed (Participants) | 219
microgram per milliliter
  Anti-1 antibody (N=219) | 2.13 [1.94 to 2.34]
  Anti-4 antibody (N=218) | 3.04 [2.77 to 3.34]
  Anti-5 antibody (N=218) | 3.24 [2.97 to 3.53]
  Anti-6B antibody (N=218) | 1.32 [1.14 to 1.54]
  Anti-7F antibody (N=218) | 3.72 [3.40 to 4.07]
  Anti-9V antibody (N=218) | 3.71 [3.37 to 4.09]
  Anti-14 antibody (N=218) | 5.27 [4.66 to 5.96]
  Anti-18C antibody (N=219) | 6.05 [5.30 to 6.89]
  Anti-19F antibody (N=219) | 5.49 [4.88 to 6.17]
  Anti-23F antibody (N=218) | 2.00 [1.70 to 2.35]

2. Primary Outcome: Antibody Concentrations Against Protein D
Description: Concentrations were given as geometric mean concentration (GMC) expressed as enzyme-linked immuno-sorbent assay (ELISA) units per milliliter.
Time Frame: One month after the administration of the 3rd vaccine dose i.e. Month 5
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: ELISA units per milliliter
Arm/Group | Synflorix Vaccine Group
Number analyzed (Participants) | 219
ELISA units per milliliter | 2923.2 [2588.6 to 3301.1]

3. Secondary Outcome: Opsonophagocytic Titer Against Pneumococcal Vaccine Serotypes
Description: The results were presented as the geometric mean dilution of serum (opsonic titer) able to sustain 50% killing of live pneumococci under the assay conditions. The vaccine pneumococcal serotypes assessed include 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F, and 23F.
Time Frame: One month after the administration of the 3rd vaccine dose i.e. Month 5
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Synflorix Vaccine Group
Number analyzed (Participants) | 97
titer
  Opsono-1 titer (N=97) | 94.1 [68.2 to 130.0]
  Opsono-4 titer (N=97) | 670.8 [516.1 to 871.7]
  Opsono-5 titer (N=94) | 148.8 [120.6 to 183.6]
  Opsono-6B titer (N=96) | 345.4 [205.5 to 580.4]
  Opsono-7F titer (N=96) | 4435.4 [3635.9 to 5410.7]
  Opsono-9V titer (N=96) | 1186.1 [955.9 to 1471.7]
  Opsono-14 titer (N=94) | 1168.3 [907.4 to 1504.2]
  Opsono-18C titer (N=94) | 222.9 [157.9 to 314.9]
  Opsono-19F titer (N=92) | 589.2 [441.9 to 785.5]
  Opsono-23F titer (N=95) | 1876.3 [1325.4 to 2656.0]

4. Secondary Outcome: Number of Subjects With Anti-pneumococcal Vaccine Serotypes Antibody Concentrations Greater Than or Equal to 0.2 Microgram Per Milliliter
Description: The vaccine pneumococcal serotypes assessed include 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F, and 23F.
Time Frame: One month after the administration of the 3rd vaccine dose i.e. Month 5
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Synflorix Vaccine Group
Number analyzed (Participants) | 219
subjects
  Anti-1 antibody (N=219) | 219
  Anti-4 antibody (N=218) | 218
  Anti-5 antibody (N=218) | 218
  Anti-6B antibody (N=218) | 203
  Anti-7F antibody (N=218) | 218
  Anti-9V antibody (N=218) | 218
  Anti-14 antibody (N=218) | 216
  Anti-18C antibody (N=219) | 218
  Anti-19F antibody (N=219) | 217
  Anti-23F antibody (N=218) | 207

5. Secondary Outcome: Antibody Concentrations Against Pneumococcal Cross-reactive Serotypes
Description: Antibody concentrations were expressed as Geometric Mean Concentrations against pneumococcal cross-reactive serotypes 6A and 19A.
Time Frame: One month after the administration of the 3rd vaccine dose i.e. Month 5
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: microgram per milliliter
Arm/Group | Synflorix Vaccine Group
Number analyzed (Participants) | 219
microgram per milliliter
  Anti-6A antibody | 0.28 [0.24 to 0.34]
  Anti-19A antibody | 0.26 [0.22 to 0.31]

6. Secondary Outcome: Opsonophagocytic Titer Against Pneumococcal Cross-reactive Serotypes
Description: The results were presented as the geometric mean dilution of serum (opsonic titer) able to sustain 50% killing of live pneumococci under the assay conditions. The cross-reactive pneumococcal serotypes assessed include 6A and 19A.
Time Frame: One month after the administration of the 3rd vaccine dose i.e. Month 5
Population: as for outcome 1
Measure: Geometric Mean (95% Confidence Interval); unit: titer
Arm/Group | Synflorix Vaccine Group
Number analyzed (Participants) | 91
titer
  Opsono-6A titer (N=91) | 159.2 [98.8 to 256.4]
  Opsono-19A titer (N=81) | 11.6 [7.3 to 18.4]

7. Secondary Outcome: Number of Subjects Seropositive Against Vaccine Pneumococcal Serotypes
Description: Seropositivity was defined as anti-pneumococcal antibody concentration greater than or equal to 0.05 microgram per milliliter. The vaccine pneumococcal serotypes assessed include 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F, and 23F.
Time Frame: One month after the administration of the 3rd vaccine dose i.e. Month 5
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Synflorix Vaccine Group
Number analyzed (Participants) | 219
subjects
  Anti-1 antibody (N=219) | 219
  Anti-4 antibody (N=218) | 218
  Anti-5 antibody (N=218) | 218
  Anti-6B antibody (N=218) | 212
  Anti-7F antibody (N=218) | 218
  Anti-9V antibody (N=218) | 218
  Anti-14 antibody (N=218) | 218
  Anti-18C antibody (N=219) | 218
  Anti-19F antibody (N=219) | 219
  Anti-23F antibody (N=218) | 212

8. Secondary Outcome: Number of Subjects Seropositive for Opsonic Titer Against Vaccine Pneumococcal Serotypes
Description: Seropositivity was defined as an opsonic titer greater than or equal to 8. The vaccine pneumococcal serotypes assessed include 1, 4, 5, 6B, 7F, 9V, 14, 18C, 19F, and 23F.
Time Frame: One month after the administration of the 3rd vaccine dose i.e. Month 5
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Synflorix Vaccine Group
Number analyzed (Participants) | 97
subjects
  Opsono-1 titer (N=97) | 83
  Opsono-4 titer (N=97) | 93
  Opsono-5 titer (N=94) | 93
  Opsono-6B titer (N=96) | 76
  Opsono-7F titer (N=96) | 96
  Opsono-9V titer (N=96) | 96
  Opsono-14 titer (N=94) | 93
  Opsono-18C titer (N=94) | 91
  Opsono-19F titer (N=92) | 90
  Opsono-23F titer (N=95) | 90

9. Secondary Outcome: Number of Subjects Seropositive Against Cross-reactive Pneumococcal Serotypes
Description: Seropositivity was defined as anti-pneumococcal antibody concentration greater than or equal to 0.05 microgram per milliliter. The cross-reactive pneumococcal serotypes assessed include 6A and 19A.
Time Frame: One month after the administration of the 3rd vaccine dose i.e. Month 5
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Synflorix Vaccine Group
Number analyzed (Participants) | 219
subjects
  Anti-6A antibody | 203
  Anti-19A antibody | 198

10. Secondary Outcome: Number of Subjects Seropositive for Opsonic Titer Against Cross-reactive Pneumococcal Serotypes
Description: Seropositivity was defined as anti-pneumococcal antibody opsonic titer greater than or equal to 8. The vaccine pneumococcal cross-reactive serotypes assessed include 6A and 19A.
Time Frame: One month after the administration of the 3rd vaccine dose i.e. Month 5
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Synflorix Vaccine Group
Number analyzed (Participants) | 91
subjects
  Opsono-6A titer (N=91) | 69
  Opsono-19A titer (N=81) | 19

11. Secondary Outcome: Number of Subjects Seropositive for Anti-Protein D Antibodies
Description: Seropositivity was defined as antibody concentration greater than or equal to 100 Enzyme-Linked Immuno Sorbent Assay (ELISA) units per milliliter.
Time Frame: One month after the administration of the 3rd vaccine dose i.e. Month 5
Population: as for outcome 1
Measure: Number; unit: subjects
Arm/Group | Synflorix Vaccine Group
Number analyzed (Participants) | 219
subjects | 219

12. Secondary Outcome: Number of Subjects Reporting Any and Grade 3 Solicited Local Adverse Events (AEs)
Description: Grade 3 redness and swelling was > 30 millimeter (mm) and grade 3 pain was subjects crying when limb was moved/spontaneously painful. Any was occurrence of any local symptom regardless of grade and whatever the number of injections.
Time Frame: Within 4 days following any vaccine dose
Population: The analysis was performed on Total Vaccinated cohort which included all subjects with the vaccine administration documented.
Measure: Number; unit: subjects
Arm/Group | Synflorix Vaccine Group
Number analyzed (Participants) | 230
subjects
  Any pain | 196
  Grade 3 pain | 80
  Any redness | 91
  Grade 3 redness | 0
  Any swelling | 178
  Grade 3 swelling | 10

13. Secondary Outcome: Number of Subjects Reporting Any, Grade 3 and Related Solicited General AEs
Description: Any fever was defined as axillary temperature ≥ 37.5 degree centigrade (°C), grade 3 fever was axillary temperature > 39.5°C. Grade 3 drowsiness, irritability, and loss of appetite was general symptom which prevented normal everyday activities. Grade 3 diarrhea was ≥ 6 looser than normal stools/day and Grade 3 vomiting was ≥ 3 episodes of vomiting/day. Related was solicited general symptom considered by the investigator to have a causal relationship to study vaccination.
Time Frame: Within 4 days following any vaccine dose
Population: as for outcome 12
Measure: Number; unit: subjects
Arm/Group | Synflorix Vaccine Group
Number analyzed (Participants) | 230
subjects
  Any diarrhea | 55
  Grade 3 diarrhea | 5
  Related diarrhea | 55
  Any drowsiness | 156
  Grade 3 drowsiness | 7
  Related drowsiness | 153
  Any fever | 147
  Grade 3 fever | 0
  Related fever | 147
  Any irritability | 198
  Grade 3 irritability | 21
  Related irritability | 196
  Any loss of appetite | 113
  Grade 3 loss of appetite | 1
  Related loss of appetite | 111
  Any vomiting | 56
  Grade 3 vomiting | 7
  Related vomiting | 56

14. Secondary Outcome: Number of Subjects Reporting Any Unsolicited AEs
Description: Unsolicited AE covers any AE reported in addition to those solicited during the clinical study and any solicited symptom with onset outside the specified period of follow-up for solicited symptoms.
Time Frame: Within 31 days after any vaccine dose
Population: as for outcome 12
Measure: Number; unit: subjects
Arm/Group | Synflorix Vaccine Group
Number analyzed (Participants) | 230
subjects | 174

15. Secondary Outcome: Number of Subjects Reporting Any Serious Adverse Events (SAEs)
Description: SAEs assessed include medical occurrences that result in death, are life threatening, require hospitalization or prolongation of hospitalization, result in disability/incapacity or are a congenital anomaly/birth defect in the offspring of a study subject.
Time Frame: Up to Month 5
Population: as for outcome 12
Measure: Number; unit: subjects
Arm/Group | Synflorix Vaccine Group
Number analyzed (Participants) | 230
subjects | 15

ADVERSE EVENTS:
Time Frame: Serious adverse events were assessed up to month 5. Systematically assessed frequent adverse events (AEs) and non-systematically assessed frequent AEs were assessed during 4 day and 31 day post vaccination period respectively.
Arm/Group | Synflorix Vaccine Group
Serious Adverse Events (participants affected / at risk) | 15/230
Other Adverse Events (participants affected / at risk) | 229/230
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix Vaccine Group (N=230)
Bronchopneumonia (Infections and infestations) | 6
Bronchiolitis (Infections and infestations) | 4
Dehydration (Metabolism and nutrition disorders) | 2
Gastroenteritis (Infections and infestations) | 2
Nasopharyngitis (Infections and infestations) | 2
Bronchial hyperreactivity (Respiratory, thoracic and mediastinal disorders) | 1
Cerebral infarction (Nervous system disorders) | 1
Conjunctivitis (Eye disorders) | 1
Convulsion (Nervous system disorders) | 1
Herpangina (Infections and infestations) | 1
Laryngitis (Infections and infestations) | 1
Pharyngitis (Infections and infestations) | 1
Pneumonia viral (Infections and infestations) | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Synflorix Vaccine Group (N=230)
Pain (General disorders) | 196
Redness (General disorders) | 91
Swelling (General disorders) | 178
Diarrhea (General disorders) | 55
Drowsiness (General disorders) | 156
Fever (General disorders) | 147
Irritability (General disorders) | 198
Loss of appetite (General disorders) | 113
Vomiting (General disorders) | 56
Nasopharyngitis (General disorders) | 123
Pharyngitis (General disorders) | 37
Conjunctivitis (General disorders) | 21
Cough (General disorders) | 17
Gastroenteritis (General disorders) | 16
Diarrhea (General disorders) | 14
Laryngitis (General disorders) | 13

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
GSK agreements may vary with individual investigators, but will not prohibit any investigator from publishing. GSK supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.